CLINICAL TRIAL: NCT02116205
Title: A Phase 2a Double-Blind, Dose-optimizing Study to Evaluate the Immunogenicity of Hantaan/Puumala Virus DNA Vaccine Administered to Healthy Adult Volunteers by Electroporation for Prevention of Hemorrhagic Fever With Renal Syndrome
Brief Title: Phase 2a Immunogenicity Study of Hantaan/Puumala Virus DNA Vaccine for Prevention of Hemorrhagic Fever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Ichor Medical Systems Incorporated (Industry); United States Army Medical Materiel Development Activity (U.S. Federal Agency); US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S-14-01; 2085 (Other: WRAIR)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Hemorrhagic Fever With Renal Syndrome
Keywords: Hantaan virus; Puumala virus; HFRS
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vaccine + Placebo at 1.0 mg (Experimental): 1.0 mg HTNV/PUUV DNA vaccine IM-EP via TriGrid™ Delivery System (TDS) on Study Day 0, 56 and 168. 1.0 mg placebo administration on Study Day 28.
  Interventions: Biological: HTNV/PUUV DNA vaccine; Biological: Placebo; Device: TriGrid Delivery System (TDS)
- Vaccine at 1.0 mg (Experimental): 1.0 mg HTNV/PUUV DNA vaccine IM-EP via TriGrid™ Delivery System (TDS) on Study Day 0, 28, 56 and 168.
  Interventions: Biological: HTNV/PUUV DNA vaccine; Device: TriGrid Delivery System (TDS)
- Vaccine + Placebo at 2.0 mg (Experimental): 2.0 mg HTNV/PUUV DNA vaccine IM-EP via TriGrid™ Delivery System (TDS) on Study Day 0, 56 and 168. 2.0 mg placebo administration on Study Day 28.
  Interventions: Biological: HTNV/PUUV DNA vaccine; Biological: Placebo; Device: TriGrid Delivery System (TDS)
- Vaccine at 2.0 mg (Experimental): 2.0 mg HTNV/PUUV DNA vaccine IM-EP via TriGrid™ Delivery System (TDS) on Study Day 0, 28, 56 and 168.
  Interventions: Biological: HTNV/PUUV DNA vaccine; Device: TriGrid Delivery System (TDS)

INTERVENTIONS:
Biological: HTNV/PUUV DNA vaccine — HTNV/PUUV DNA vaccine mixture, composed of pWRG/HTN-M(co) and pWRG/PUU-M(s2)
  Other Names: Hantaan Virus/Puumala Virus DNA Vaccine
Biological: Placebo — 0.9% sodium chloride
  Other Names: Normal saline placebo
  Arms: Vaccine + Placebo at 1.0 mg; Vaccine + Placebo at 2.0 mg
Device: TriGrid Delivery System (TDS) — The TDS-IM is an integrated, fully automated clinical EP system designed for delivering DNA-based vaccines and therapies to target tissues, through temporary disruption of cellular membranes via electrical pulses
  Other Names: TriGrid Delivery System for intramuscular delivery (TDS-IM)

SUMMARY:
The purpose of this study is to compare the immune responses of two different doses (1.0 mg and 2.0 mg) and two different dosing schedules (two doses or three doses) of a mixed Hantaan virus (HTNV) and Puumala virus (PUUV) DNA vaccine in healthy participants. To maintain a blind, participants in the two-dose group will receive one dose of normal saline placebo. All of the groups will also receive a booster dose 6 months after first vaccination. The results will help to determine which dose and vaccination schedule will be best to move forward in the vaccine development process.

DETAILED DESCRIPTION:
The study will enroll 4 randomized groups of 30 subjects each for a total of 120 subjects. These groups will be split so that 60 individuals receive the 1.0 mg dose and the other 60 receive the 2.0 mg dose. Every subject will receive a total of 3 injections on Days 0, 28, and 56. Half of each of these groups (n = 30) will receive 2 vaccine injections at Days 0 and 56 (normal saline placebo on Day 28) while the other half will receive 3 vaccine injections at Days 0, 28, and 56. All subjects will receive a booster dose at Day 168 to help assess immunogenicity with this booster dose. All doses will be administered with the TDS-IM device. All subjects will be followed until at least Day 252 (a 12 month follow-up visit may be requested). Subjects will complete post-injection memory aids for 7 days after each injection. There will also be up to 12 alternates enrolled and used to replace any original subject who fails to complete all 3 scheduled primary injections and Day 70 follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-pregnant, non-lactating female, ages 18-49 (inclusive) at the time of screening
* Have provided written informed consent before screening
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination prior to entry into the study
* Available and able to participate for all study visits and procedures
* Females, if sexually active, are known to be at least one year post-menopausal (defined as no menses for 12 consecutive months), or willing to use an effective method of contraception (eg, hormonal contraception, diaphragm, cervical cap, intrauterine device, condom, anatomical sterility [self or partner]) from the date of screening until at least 3 months after the last injection
* Negative hantavirus pseudovirion neutralization assay (PsVNA) test result at screening

Exclusion Criteria:

* History or serologic evidence of prior infection with any hantavirus virus, or prior participation in a HTNV or PUUV vaccine trial
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* Ongoing participation in another clinical trial
* Receipt or planned receipt of any vaccination, experimental or otherwise within the period 30 days prior to the first injection through the period 60 days after Study Day 168 (booster dose; approximately 9 month period in total), with the exception of emergency use vaccinations as needed
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for all eligible injection sites (deltoid region) exceeds 40 mm
* Individuals in whom the ability to observe possible local reactions at the eligible injections sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical exam, electrocardiogram (ECG), and/or laboratory screening test
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* Any serologic evidence of hepatitis B or C infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of study entry

  1. For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day
  2. Intranasal and topical steroids are allowed
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child
* Syncopal episode within 12 months of screening
* Suspected or known current alcohol and/or illicit drug abuse
* Unwilling to allow storage and use of blood for future hantavirus-related research
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher Paolino, MD, Principal Investigator — WRAIR Clinical Trials Center
Locations (1):
- Walter Reed Army Institute of Research Clinical Trials Center, Silver Spring, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 130 subjects were enrolled in the study. Ten of the 130 were enrolled as replacements for early withdrawals. The first participant was enrolled on July 9, 2014 and the last participant was enrolled in September 2015.
Period: Overall Study
Arm/Group | Vaccine + Placebo at 1.0 mg | Vaccine at 1.0 mg | Vaccine + Placebo at 2.0 mg | Vaccine at 2.0 mg
Started | 31 | 33 | 33 | 33
Completed | 29 | 26 | 29 | 27
Not Completed | 2 | 7 | 4 | 6
Not completed — Withdrawal by Subject | 2 | 4 | 1 | 3
Not completed — Lost to Follow-up | 0 | 2 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 1
Not completed — Exclusion criteria | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine + Placebo at 1.0 mg | Vaccine at 1.0 mg | Vaccine + Placebo at 2.0 mg | Vaccine at 2.0 mg | Total
Number analyzed (Participants) | 31 | 33 | 33 | 33 | 130
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 34.3 (8.8) | 30.9 (8.9) | 30.5 (6.6) | 33.2 (8.5) | 32.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 13 | 18 | 63
  Male | 16 | 16 | 20 | 15 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 3 | 1 | 11
  Not Hispanic or Latino | 29 | 28 | 30 | 32 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 20 | 17 | 14 | 15 | 66
  White | 11 | 13 | 14 | 13 | 51
  More than one race | 0 | 1 | 2 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 33 | 33 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroconversion of HTNV and PUUV Using PsVNA50
Description: The primary endpoint will be to determine the seroconversion rates of the vaccines. Seroconversion is defined as production of neutralizing antibody titers measured using a pseudovirion neutralization assay (PsVNA). A PsVNA50 titer ≥ 20 is considered positive. Sera were collected on Days 0, 28, 56, 84, 140, 168, 196, 252, 365 and evaluated for the presence of neutralizing antibodies using PsVNA50. Percentages for seroconversion are based on the number of subjects presenting non-missing data.
Time Frame: Study Days 0 to 365
Population: Of the 130 subjects enrolled, 120 met the conditions for the efficacy evaluable population, that is subjects who received all three of the vaccinations on Study Days 0, 28, and 56; and who attended at least one subsequent study visit. Seroconversion is measured in the efficacy evaluable population.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine + Placebo at 1.0 mg | Vaccine at 1.0 mg | Vaccine + Placebo at 2.0 mg | Vaccine at 2.0 mg
Number analyzed (Participants) | 30 | 30 | 30 | 30
Participants
  Seroconversion at Day 28: Seroconversion | 1 | 1 | 1 | 2
  Seroconversion at Day 28: No Seroconversion | 29 | 29 | 29 | 28
  Seroconversion at Day 56: Seroconversion | 1 | 10 | 1 | 7
  Seroconversion at Day 56: No Seroconversion | 29 | 20 | 29 | 23
  Seroconversion at Day 84: Seroconversion | 15 | 18 | 14 | 17
  Seroconversion at Day 84: No Seroconversion | 15 | 12 | 16 | 13
  Seroconversion at Day 140: number analyzed (Participants) | 30 | 28 | 29 | 28
  Seroconversion at Day 140: Seroconversion | 11 | 14 | 9 | 12
  Seroconversion at Day 140: No Seroconversion | 19 | 14 | 20 | 16
  Seroconversion at Day 168: number analyzed (Participants) | 30 | 27 | 29 | 26
  Seroconversion at Day 168: Seroconversion | 12 | 11 | 7 | 13
  Seroconversion at Day 168: No Seroconversion | 18 | 16 | 22 | 13
  Seroconversion at Day 196: number analyzed (Participants) | 30 | 26 | 29 | 27
  Seroconversion at Day 196: Seroconversion | 18 | 23 | 20 | 19
  Seroconversion at Day 196: No Seroconversion | 12 | 3 | 9 | 8
  Seroconversion at Day 252: number analyzed (Participants) | 29 | 26 | 29 | 27
  Seroconversion at Day 252: Seroconversion | 12 | 16 | 19 | 16
  Seroconversion at Day 252: No Seroconversion | 17 | 10 | 10 | 11
  Seroconversion at Day 365: number analyzed (Participants) | 20 | 22 | 22 | 20
  Seroconversion at Day 365: Seroconversion | 12 | 15 | 16 | 14
  Seroconversion at Day 365: No Seroconversion | 8 | 7 | 6 | 6

2. Secondary Outcome: Number of Solicited Adverse Events (AEs) in Study Subjects
Description: The nature, frequency, and severity of solicited adverse events (AE) occurring from the time of each injection through 14 days following the procedure. The total number of events counts all solicited adverse events for all subjects. Subjects may have more than one solicited adverse event per body system and preferred term.
Time Frame: The time of each injection through 14 days following the procedure
Measure: Number; unit: Adverse Events
Arm/Group | Vaccine + Placebo at 1.0 mg | Vaccine at 1.0 mg | Vaccine + Placebo at 2.0 mg | Vaccine at 2.0 mg
Number analyzed (Participants) | 31 | 33 | 33 | 33
Adverse Events
  Total Number of Events | 144 | 148 | 173 | 182
  Mild | 131 | 136 | 147 | 155
  Moderate | 13 | 9 | 25 | 24
  Severe | 0 | 3 | 1 | 3
  Life Threatening | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Seroconversion of HTNV and PUUV Using PsVNA80
Description: Seroconversion is defined as production of neutralizing antibody titers measured using a pseudovirion neutralization assay (PsVNA). Sera were collected on Days 0, 28, 56, 84, 140, 168, 196, 252, 365 and evaluated for the presence of neutralizing antibodies by using PsVNA80. Percentages for seroconversion are based on the number of subjects presenting non-missing data.
Time Frame: Study Days 0 to 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine + Placebo at 1.0 mg | Vaccine at 1.0 mg | Vaccine + Placebo at 2.0 mg | Vaccine at 2.0 mg
Number analyzed (Participants) | 30 | 30 | 30 | 30
Participants
  Seroconversion at Day 28: Seroconversion | 0 | 1 | 0 | 2
  Seroconversion at Day 28: No Seroconversion | 30 | 29 | 30 | 28
  Seroconversion at Day 56: Seroconversion | 0 | 6 | 0 | 1
  Seroconversion at Day 56: No Seroconversion | 30 | 24 | 30 | 29
  Seroconversion at Day 84: Seroconversion | 5 | 13 | 8 | 9
  Seroconversion at Day 84: No Seroconversion | 25 | 17 | 22 | 21
  Seroconversion at Day 140: number analyzed (Participants) | 30 | 28 | 29 | 28
  Seroconversion at Day 140: Seroconversion | 2 | 8 | 4 | 5
  Seroconversion at Day 140: No Seroconversion | 28 | 20 | 25 | 23
  Seroconversion at Day 168: number analyzed (Participants) | 30 | 27 | 29 | 26
  Seroconversion at Day 168: Seroconversion | 4 | 8 | 3 | 3
  Seroconversion at Day 168: No Seroconversion | 26 | 19 | 26 | 23
  Seroconversion at Day 196: number analyzed (Participants) | 30 | 26 | 29 | 27
  Seroconversion at Day 196: Seroconversion | 14 | 19 | 17 | 16
  Seroconversion at Day 196: No Seroconversion | 16 | 7 | 12 | 11
  Seroconversion at Day 252: number analyzed (Participants) | 29 | 26 | 29 | 27
  Seroconversion at Day 252: Seroconversion | 6 | 13 | 9 | 10
  Seroconversion at Day 252: No Seroconversion | 23 | 13 | 20 | 17
  Seroconversion at Day 365: number analyzed (Participants) | 20 | 22 | 22 | 20
  Seroconversion at Day 365: Seroconversion | 5 | 9 | 4 | 9
  Seroconversion at Day 365: No Seroconversion | 15 | 13 | 18 | 11

ADVERSE EVENTS:
Time Frame: Study Days 0 to 365
Description: Solicited and unsolicited adverse events for all subjects who received at least one dose of vaccine reported
Arm/Group | Vaccine + Placebo at 1.0 mg | Vaccine at 1.0 mg | Vaccine + Placebo at 2.0 mg | Vaccine at 2.0 mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33 | 1/33 | 0/33
Other Adverse Events (participants affected / at risk) | 29/31 | 33/33 | 31/33 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine + Placebo at 1.0 mg (N=31) | Vaccine at 1.0 mg (N=33) | Vaccine + Placebo at 2.0 mg (N=33) | Vaccine at 2.0 mg (N=33)
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Enteritis vs Alcohol Induced Gastritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine + Placebo at 1.0 mg (N=31) | Vaccine at 1.0 mg (N=33) | Vaccine + Placebo at 2.0 mg (N=33) | Vaccine at 2.0 mg (N=33)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 3 | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Axillary pain (General disorders) | 2 | 2 | 4 | 4
Fatigue (General disorders) | 9 | 4 | 13 | 12
Injection site bruising (General disorders) | 3 | 2 | 1 | 3
Injection site erythema (General disorders) | 3 | 3 | 6 | 6
Injection site pain (General disorders) | 29 | 33 | 30 | 33
Injection site reaction (General disorders) | 1 | 4 | 4 | 2
Injection site swelling (General disorders) | 1 | 1 | 0 | 2
Local swelling (General disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Respiratory rate increased (Investigations) | 1 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 8 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 7 | 7 | 9 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Scleral discolouration (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 1 | 2
Allergy to chemicals (Immune system disorders) | 0 | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 1 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 7 | 10
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0
Blood pressure diastolic increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Grip strength decreased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 5 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Libido increased (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No